CLINICAL TRIAL: NCT02674230
Title: OCEAN Registry: Obesity and Clock for Elegant Aging Registry 肥胖控制及生理時鐘之研究計畫
Brief Title: OCEAN Registry: Obesity and Clock for Elegant Aging Registry
Acronym: OCEAN
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chao-Yung Wang, Doctor, Chang Gung Memorial Hospital
Other Study IDs: 100-0250A3
Record Dates: First submitted 2016-01-26; First posted 2016-02-04 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Circadian Dysregulation; Aging; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Chronobiology Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — A. Serum. B. White blood cells. C. Adipose tissue. (If receiving liposuction, plastic surgery, bariatric surgery, dermatological procedure, intra-abdominal operation, and cardiovascular surgery)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Extreme obesity: BMI ≥35kg/m2
- Obesity: BMI 24-34.9kg/m2
- Normal subjects: BMI <24kg/m2. No systemic disease, including hypertension, diabetes, liver cirrhosis, chronic kidney disease, and psychiatric disease.

SUMMARY:
This study aims to study the relationships between obesity, circadian rhythm, and aging. The investigators set up a prospective cohort registry for morbid obesity, obesity, and normal subjects with annual follow-up. The cohort aims to investigate the pathophysiological, molecular, genetic, and cellular aspects of the relationships between obesity, circadian deregulation, and impacts on aging. Clinical data, questionnaires, biological material, and molecular signatures will be collected and investigated.

DETAILED DESCRIPTION:
The objective of this observational study is the follow-up of 2000 adult obesity (BMI ≥ 35 and 24-35 kg/m2) and non-obese subjects with annual follow-up for 10 years. Clinical data, biochemistry, and biological samples (serum, DNA, RNA, white blood cells) will be collected and stored. Adipose tissues will be collected if participants received liposuction, plastic surgery, bariatric surgery, dermatological procedure, intra-abdominal operation, and cardiovascular surgery. Questionnaires will be obtained with special nurse including sleep quality, chronotypes, and circadian activities. During follow up period, major adverse cardiovascular events will be monitored.

The investigators anticipate that the results generated from the study will provide valuable data to a better understanding of the relationships between obesity, circadian rhythm, and aging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Body mass index ≥ 24 kg/m2
* For normal subjects, Body mass index < 24 kg/m2

Exclusion Criteria:

* No inform consent
* Use of steroid medications
* Severe systemic diseases or organ failure with estimated life expectancy of 6 months or less

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the general population including healthcare facility and non-health care settings. Healthcare facility includes university based hospital and primary care clinics. Non-health care settings include schools, subjects families, and employment agencies.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-07; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Body weight | 10 years

SECONDARY OUTCOMES:
Major Cardiovascular Adverse Events | 3, 6, 12, and 18 months. 2, 5, and 10 years
Sleep quality as assessed by Pittsburgh Sleep Quality Index (PSQI) questionnaire | 3, 6, 12, and 18 months. 2, 5, and 10 years
Personal chronotype (biological clock) as assessed by Munich Chronotype Questionnaire | 3, 6, 12, and 18 months. 2, 5, and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Yung Wang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided